CLINICAL TRIAL: NCT01632995
Title: Implementation of HIV Pre-exposure Prophylaxis (PrEP): A Demonstration Project
Brief Title: Assessment of Pre-Exposure Prophylaxis (PrEP) Administered at Sexually Transmitted Disease (STD) Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PrEP Demonstration Project; 11879 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2016-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Racivir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

ARMS (1):
- Emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) (Experimental): All study participants will be assigned to this arm and will receive one FTC/TDF tablet orally once a day.
  Interventions: Drug: FTC 200 mg/TDF 300 mg fixed-dose combination tablet

INTERVENTIONS:
Drug: FTC 200 mg/TDF 300 mg fixed-dose combination tablet — Each participant will be directed to take one FTC/TDF tablet orally once a day, with or without food.
  Other Names: Truvada

SUMMARY:
This study will assess the uptake, acceptability, safety, and feasibility of HIV pre-exposure prophylaxis (PrEP), consisting of a once-daily fixed-dose combination tablet of emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF), administered at sexually transmitted disease (STD) clinics and a community health center in the United States.

DETAILED DESCRIPTION:
A previous study (iPrEx) showed that daily PrEP with FTC/TDF provided with a comprehensive package of prevention services is effective in preventing HIV infection among men who have sex with men (MSM). The PrEP administered in that study was given in the context of a research setting/controlled trial, but it is important to evaluate the acceptability, sustainability, and safety of PrEP in a "real world" setting. This study will evaluate PrEP administered to HIV-uninfected MSM and transgender females at two STD clinics and one community health center in the United States.

Each participant will receive PrEP for up to 1 year and will have up to 8 study visits. PrEP will consist of one fixed-dose FTC/TDF combination tablet orally each day. All participants will have study visits at screening, enrollment, and 4 weeks after enrollment; participants will continue to have visits at Weeks 12, 24, 36, 48, and 52 if they do not seroconvert. Participants who seroconvert will discontinue PrEP and will have a post-drug discontinuation visit 4 weeks after discontinuing PrEP. At most visits, participants will undergo blood, urine, and hair sample collection; give a medical history; undergo a physical exam; receive risk-reduction counseling and condoms; undergo testing for HIV and other STDs; receive study drugs; and undergo a pill count and adherence assessment (follow-up visits only). For participants who stop taking the study drug but remain in the study, urine, blood, and hair samples will not be collected at 12-week follow-up visits if all stop procedures have been completed and if there are no lab abnormalities that require additional follow-up. Participants will also answer questionnaires at screening, 12-week visits, and at study exit.

ELIGIBILITY:
Inclusion Criteria:

* Must be either a man who has sex with men or a transgender female
* Male sex (at birth)
* Willing and able to provide written informed consent
* HIV-1 uninfected, defined as having a negative rapid HIV antibody test at both screening visit and enrollment and a negative 4th generation antibody/antigen test at screening
* No laboratory evidence of a detectable HIV viral load (San Francisco site only)
* Evidence of risk of acquiring HIV-1 infection including any one of the following:

  (1) Condomless anal sex with two or more male or transgender female sex partners during the last 12 months; or (2) two or more episodes of anal sex with at least one HIV-positive partner during the last 12 months; or (3) sex with a male or transgender female partner and any of the following STDs diagnosed during the last 12 months or at screening: syphilis, rectal gonorrhea, or rectal chlamydia.
* Able to provide a street address of residence or phone number for themselves or two personal contacts who would know their whereabouts during the period of the demonstration project
* Adequate renal function: creatinine clearance of 60 ml/min or greater as estimated by the Cockcroft-Gault equation within 45 days of enrollment
* A urine dipstick with a negative or trace result for protein within 45 days of enrollment
* Fluent in English or in Spanish

Exclusion Criteria:

* Signs or symptoms of acute HIV infection
* Previously diagnosed active and serious infections including active tuberculosis infection or osteomyelitis and all infections requiring parenteral antibiotic therapy (other than STDs requiring intramuscular injections of antibiotics); active clinically significant medical problems including poorly controlled cardiac disease (e.g., symptoms of ischemia or congestive heart failure) or previously diagnosed malignancy expected to require further treatment
* Hepatitis B surface antigen (HBsAg) positive
* History of pathological bone fractures not related to trauma
* Receiving ongoing therapy with any of the following: investigational antiretroviral agents (PEP is allowed as described in the protocol), interferon (alpha, beta, or gamma) or interleukin (e.g., IL-2) therapy, agents with significant nephrotoxic potential, other agents that may inhibit or compete for elimination via active renal tubular secretion (e.g., probenecid), and/or other investigational agents
* Concomitant participation in a clinical trial using investigational agents, including placebo-controlled clinical trials using such agents
* At enrollment, has any other condition that, based on the opinion of the investigator or designee, would preclude provision of informed consent; make participation in the project unsafe; complicate interpretation of outcome data; or otherwise interfere with achieving the project objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2012-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Liu, MD, MPH, Study Chair — San Francisco Department of Public Health
Locations (3):
- United States (3):
  - SF City Clinic Non-Network CRS, San Francisco, California
  - Whitman Walker Non-network CRS, Washington D.C., District of Columbia
  - Miami PrEP Non-Network CRS, Miami, Florida

REFERENCES:
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and enrolled at 3 sites in the US (San Francisco, Miami, Washington DC). Enrollment began on October 1, 2012 and ended February 10, 2015.
Pre-assignment Details: As this PrEP Demonstration project assessed acceptance of PrEP, all participants assessed for participation are included in the "start" category, and those who enrolled and initiated PrEP are indicated as a separate milestone.
Period: Pre-screening to Enrollment Period
Arm/Group | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF)
Started (All participants who were assessed for study participation) | 1069
Completed (All participants who enrolled in study) | 557
Not Completed | 512
Period: Main Study Follow-up Period
Arm/Group | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF)
Started (Participants who enrolled and initiated PrEP) | 557
Completed (Participants who completed 48 weeks of follow-up) | 437
Not Completed | 120

BASELINE CHARACTERISTICS:
Arm/Group | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF)
Number analyzed (Participants) | 557
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [27 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 557
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 266
  Latino | 192
  Black | 40
  Asian | 26
  Other | 32
Region of Enrollment [Number; unit: participants]
  United States | 557

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Acceptance Rate of PrEP
Time Frame: Measured through enrollment (Week 0)
Measure: Count of Participants; unit: Participants
Groups:
- Participants Assessed for Participation: All participants who were assessed for study participation
Arm/Group | Participants Assessed for Participation
Number analyzed (Participants) | 1069
Participants
  Potentially eligible clients | 921
  Participants enrolled | 557

2. Primary Outcome: Measurement of Refusal Rate of PrEP
Time Frame: Measured through enrollment (Week 0)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Assessed for Participation
Number analyzed (Participants) | 1069
Participants
  Potentially eligible clients | 921
  Declined participation | 364

3. Primary Outcome: Duration of PrEP Use
Description: Number of study drug interruptions
Time Frame: Participants were followed for 48 weeks, or up to the point of early termination
Measure: Number; unit: interruptions
Arm/Group | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF)
Number analyzed (Participants) | 557
interruptions | 86

4. Primary Outcome: Duration of PrEP Use
Description: Mean duration of interruptions
Time Frame: Participants were followed for 48 weeks, or up to the point of early termination
Measure: Number; unit: Days
Arm/Group | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF)
Number analyzed (Participants) | 557
Days | 65

5. Primary Outcome: Measurement of Side Effects/Toxicities
Time Frame: Participants were followed for 48 weeks, or up to the point of early termination
Measure: Number; unit: events
Arm/Group | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF)
Number analyzed (Participants) | 557
events
  Serious adverse events | 19
  Creatinine elevations | 23

6. Primary Outcome: Measurement of PrEP Adherence by TFV-DP Levels in DBS
Time Frame: Participants were followed for 48 weeks, or up to the point of early termination
Population: DBS testing was performed in approximately 100 randomly selected participants per site, and among all African American and transgender participants, who were underrepresented in the overall sample
Measure: Number; unit: Percent of Participants
Groups:
- Participants With DBS Testing: All study participants who had at least 1 DBS result
Arm/Group | Participants With DBS Testing
Number analyzed (Participants) | 294
Percent of Participants
  % with protective TFV-DP levels at week 4 | 86
  % with protective TFV-DP levels at week 12 | 85
  % with protective TFV-DP levels at week 24 | 82
  % with protective TFV-DP levels at week 36 | 85
  % with protective TFV-DP levels at week 48 | 80

7. Primary Outcome: Number of Male Sexual Partners
Time Frame: Participants were followed for 48 weeks, or up to the point of early termination
Measure: Mean (Full Range); unit: partners
Arm/Group | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF)
Number analyzed (Participants) | 557
partners
  Mean Anal sex partners at baseline | 10.9 [0 to 120]
  Mean Anal sex partners at week 48 | 9.3 [0 to 240]

8. Primary Outcome: Measurement of PrEP Adherence by Medication Possession Ratio
Description: Medication possession ratio is defined as the number of dispensed pills divided by the number of days between visits
Time Frame: Participants were followed for 48 weeks, or up to the point of early termination
Population: Mean PrEP adherence by medication possession ratio
Measure: Number; unit: percent
Arm/Group | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF)
Number analyzed (Participants) | 557
percent | 85.9

9. Secondary Outcome: Number of Participants Who Seroconvert
Time Frame: Participants were followed for 48 weeks, or up to the point of early termination
Measure: Number; unit: participants
Arm/Group | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF)
Number analyzed (Participants) | 557
participants
  Acute HIV infection at baseline | 3
  HIV seroconversion during follow-up | 2

10. Secondary Outcome: Measurement of HIV Drug Resistance Patterns Among Participants Who Become Infected
Time Frame: Participants were followed for 48 weeks, or up to the point of early termination
Measure: Number; unit: participant with acquired HIV resistance
Arm/Group | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF)
Number analyzed (Participants) | 557
participant with acquired HIV resistance | 1

ADVERSE EVENTS:
Arm/Group | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF)
Serious Adverse Events (participants affected / at risk) | 19/557
Other Adverse Events (participants affected / at risk) | 25/557
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF) (N=557)
suicidal ideation and/or attempt, bipolar disorder, or anxiety (Psychiatric disorders) | 8 (8) — Assessed as not related to study drug
Hypertension / Hypertensive crisis (General disorders) | 2 (2)
Appendicitis (Gastrointestinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Testicular torsion (Injury, poisoning and procedural complications) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Food allergy (Immune system disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emtricitabine (FTC)/Tenofovir Disoproxil Fumarate (TDF) (N=557)
Creatinine elevation (Investigations) | 13 (23)
Bone fracture (Injury, poisoning and procedural complications) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No